CLINICAL TRIAL: NCT03481634
Title: A Two-year, Three-arm, Randomized, Double-masked, Multicenter, Phase III Study Assessing the Efficacy and Safety of Brolucizumab Versus Aflibercept in Adult Patients With Visual Impairment Due to Diabetic Macular Edema
Brief Title: Study of Efficacy and Safety of Brolucizumab vs. Aflibercept in Patients With Visual Impairment Due to Diabetic Macular Edema
Acronym: KESTREL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRTH258B2301; 2017-004742-23 (EudraCT Number)
Record Dates: First submitted 2018-03-13; First posted 2018-03-29 (Actual); Results first posted 2022-10-28 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; intravitreal injection; brolucizumab; aflibercept; double-masked; Diabetic Macular Edema (DME); macular edema; diabetic retinopathy
MeSH Terms: conditions — Macular Edema; Diabetic Retinopathy | interventions — brolucizumab; aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Brolucizumab 3 mg (Experimental): Brolucizumab 3 mg/0.05 mL, 5 loading doses, with subsequent doses per protocol-specified maintenance schedule.
  To fulfil the double-masking requirement, each investigational site had masked and unmasked staff. The investigator who performed the injection was unmasked to the treatments as were any other site personnel who had been delegated responsibility for working with the Investigational Product (IP).
  Interventions: Drug: Brolucizumab
- Brolucizumab 6 mg (Experimental): Brolucizumab 6 mg/0.05 mL, 5 loading doses, with subsequent doses per protocol-specified maintenance schedule.
  To fulfil the double-masking requirement, each investigational site had masked and unmasked staff. The investigator who performed the injection was unmasked to the treatments as were any other site personnel who had been delegated responsibility for working with the Investigational Product (IP).
  Interventions: Drug: Brolucizumab
- Aflibercept 2 mg (Active Comparator): Aflibercept 2 mg/0.05 mL, as labeled, 5 loading doses, with subsequent doses every 8 weeks.
  To fulfil the double-masking requirement, each investigational site had masked and unmasked staff. The investigator who performed the injection was unmasked to the treatments as were any other site personnel who had been delegated responsibility for working with the Investigational Product (IP).
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Brolucizumab — Intravitreal injection
  Other Names: RTH258; ESBA1008
  Arms: Brolucizumab 3 mg; Brolucizumab 6 mg
Drug: Aflibercept — Intravitreal injection
  Other Names: Eylea
  Arms: Aflibercept 2 mg

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of brolucizumab in treatment of patients with visual impairment due to diabetic macular edema (DME).

DETAILED DESCRIPTION:
This was a Phase III, randomized, double-masked, multi-center, active-controlled, three-arm study designed to evaluate the efficacy and safety of brolucizumab 6 mg and 3 mg compared to the active control, aflibercept 2 mg used per authorized label, in subjects with diabetic macular edema (DME). The study included a screening period of up to 2 weeks to assess eligibility, followed by a doublemasked treatment period (Day 1 to Week 96). The baseline visit was defined as Day 1/Visit 1, and end of treatment visit as Visit 27 (Week 96). After the last treatment visit, a post-treatment follow-up period was planned from Week 96 to Week 100.

Subjects were assigned to one of three treatment arms in a 1:1:1 ratio: brolucizumab 6 mg/0.05 mL administered 5 x every 6 weeks (q6w) during loading phase then q12w/every 8 weeks (q8w) during maintenance phase, brolucizumab 3 mg/0.05 mL administered 5 x every 6 weeks (q6w) during loading phase then q12w/q8w during maintenance phase or aflibercept 2 mg/0.05 mL administered 5 x every 4 weeks (q4w) during loading phase then q8w during maintenance phase.

Disease Activity Assessments (DAAs) were conducted by the masked investigator for each treatment arm at Week 32 and Week 36, i.e. 8 and 12 weeks after the end of the loading phase for subjects receiving brolucizumab. Assessments were also performed at Week 48, and will then continue to be performed from Week 60 up to Week 96, every 12 weeks. Subjects in the brolucizumab arms who qualified for q12w during the initial q12w interval continued on a q12w treatment frequency unless disease activity was identified at any of the subsequent DAA visits, in which case subjects were switched to a q8w treatment interval until the end of the study.

To fulfil the double-masking requirement, each investigational site had masked and unmasked staff. The investigator who performed the injection was unmasked to the treatments as were any other site personnel who had been delegated responsibility for working with the Investigational Product (IP). The unmasked site personnel and unmasked injecting investigator did not perform Best-corrected visual acuity (BCVA), complete ophthalmic examination (with the exception of post-injection safety assessment), DAAs or administer the Visual Functioning Questionnaire-25 (VFQ-25). Also, the unmasked site personnel and unmasked injecting physician did not perform assessment of any ocular or non-ocular safety parameters, or assess causality of Adverse event (AEs) for subjects during the course of the study except an event reported immediately following Intravitreal treatment (IVT). Once the designated roles were determined, the unmasked investigator/site personnel roles were not switched at any time after randomization to masked role. Every effort was made to limit the number of unmasked study personnel to ensure the integrity of this masked study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent before any assessment
* Patients with type 1 or type 2 diabetes mellitus and HbA1c of ≤10% at screening
* Medication for the management of diabetes stable within 3 months prior to randomization and is expected to remain stable during the course of the study

Exclusion Criteria:

* Active proliferative diabetic retinopathy in the study eye
* Active intraocular or periocular infection or active intraocular inflammation in study eye
* Uncontrolled glaucoma in the study eye defined as intraocular pressure (IOP) > 25 millimeters mercury (mmHg)
* Previous treatment with anti-VEGF drugs or investigational drugs in the study eye
* Stroke or myocardial infarction during the 6-month period prior to baseline
* Uncontrolled blood pressure defined as a systolic value ≥160 mmHg or diastolic value ≥100 mmHg

Other protocol-specified inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 566 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2021-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (102):
- United States (36):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, La Jolla, California
  - Novartis Investigative Site, Mountain View, California
  - Novartis Investigative Site, Santa Barbara, California
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Danbury, Connecticut
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Pensacola, Florida
  - Novartis Investigative Site, Stuart, Florida
  - Novartis Investigative Site, ‘Aiea, Hawaii
  - Novartis Investigative Site, Urbana, Illinois
  - Novartis Investigative Site, Wheaton, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, New Albany, Indiana
  - Novartis Investigative Site, Leawood, Kansas
  - Novartis Investigative Site, Lenexa, Kansas
  - Novartis Investigative Site, Paducah, Kentucky
  - Novartis Investigative Site, Springfield, Massachusetts
  - Novartis Investigative Site, Stoneham, Massachusetts
  - Novartis Investigative Site, Reno, Nevada
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Kingston, Pennsylvania
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Memphis, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Bellaire, Texas
  - Novartis Investigative Site, Harlingen, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Tyler, Texas
  - Novartis Investigative Site, Silverdale, Washington
  - Novartis Investigative Site, Spokane, Washington
  - Novartis Investigative Site, Madison, Wisconsin
- Argentina (4):
  - Novartis Investigative Site, Ciudad Autonoma de Bs As, Buenos Aires
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, CABA
  - Novartis Investigative Site, Córdoba
- Australia (8):
  - Novartis Investigative Site, Liverpool, New South Wales
  - Novartis Investigative Site, Parramatta, New South Wales
  - Novartis Investigative Site, Sydney, New South Wales
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
- Austria (3):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Vienna
- Canada (3):
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Québec
- Colombia (2):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Bogotá
- Israel (6):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Rehovot
  - Novartis Investigative Site, Tel Aviv
- Italy (5):
  - Novartis Investigative Site, Chieti, CH
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Roma, RM
- Japan (15):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Amagasaki, Hyōgo
  - Novartis Investigative Site, Tsuchiura, Ibaragi
  - Novartis Investigative Site, Ishioka, Ibaraki
  - Novartis Investigative Site, Kagoshima, Kagoshima-ken
  - Novartis Investigative Site, Matsumoto, Nagano
  - Novartis Investigative Site, Saitama-shi, Saitama
  - Novartis Investigative Site, Shimotsuke, Tochigi
  - Novartis Investigative Site, Chiyoda-ku, Tokyo
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Taito-ku, Tokyo
  - Novartis Investigative Site, Kumamoto
  - Novartis Investigative Site, Osaka
- Netherlands (3):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, Tilburg
- Portugal (5):
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Leiria
  - Novartis Investigative Site, Porto
  - Novartis Investigative Site, Santa Maria da Feira
  - Novartis Investigative Site, Vila Franca de Xira
- Novartis Investigative Site, Arecibo, Puerto Rico
- Spain (6):
  - Novartis Investigative Site, Valladolid, Castille and León
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Sant Cugat del Vallès, Catalonia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Zaragoza
- United Kingdom (5):
  - Novartis Investigative Site, Frimley, Surrey
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Hull
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1194

RESULTS

PARTICIPANT FLOW:
Groups:
- Brolucizumab 3 mg: Brolucizumab 3 mg/0.05 mL, 5 loading doses, with subsequent doses per protocol-specified maintenance schedule
- Brolucizumab 6 mg: Brolucizumab 6 mg/0.05 mL, 5 loading doses, with subsequent doses per protocol-specified maintenance schedule
- Aflibercept 2 mg: Aflibercept 2 mg/0.05 mL, as labeled, 5 loading doses, with subsequent doses every 8 weeks
Period: Overall Study
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Started | 190 | 189 | 187
Completed | 157 | 154 | 153
Not Completed | 33 | 35 | 34
Not completed — Withdrawal by Subject | 16 | 19 | 14
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Progressive disease | 0 | 1 | 0
Not completed — Physician Decision | 3 | 0 | 1
Not completed — Lost to Follow-up | 3 | 4 | 4
Not completed — Death | 4 | 8 | 7
Not completed — Adverse Event | 6 | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg | Total
Number analyzed (Participants) | 190 | 189 | 187 | 566
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 97 | 104 | 93 | 294
  >=65 years | 93 | 85 | 94 | 272
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (9.76) | 62.4 (10.14) | 63.9 (10.09) | 63.6 (10.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 79 | 61 | 211
  Male | 119 | 110 | 126 | 355
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 25 | 25 | 26 | 76
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 2
  Black or African American | 13 | 4 | 7 | 24
  White | 151 | 158 | 152 | 461
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best-corrected Visual Acuity (BCVA) at Week 52
Description: BCVA was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts.
  Visual Function of the study eye was assessed using the ETDRS protocol. Participants with a BCVA ETDRS letter score of 78 to 23 (approximate Snellen equivalent of 20/32 to 20/320) in the study eye were included.
  Min and max possible scores are 0-100 respectively. A higher score represents better visual functioning.
  This endpoint was analyzed via the pairwise ANOVA method where the 2 dose groups of Brolucizumab are compared to Aflibercept.
Time Frame: Baseline, Week 52
Population: Full analysis set (FAS) - Last observation carried forward (LOCF).
  This endpoint was analyzed via the pairwise ANOVA method where the 2 dose groups of Brolucizumab are compared to Aflibercept
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 190 | 189 | 187
Scores on a scale
  LS mean estimate (Brolucizumab 3 mg vs. Aflibercept 2 mg): number analyzed (Participants) | 190 | 0 | 187
  LS mean estimate (Brolucizumab 3 mg vs. Aflibercept 2 mg) | 7.3 (0.66) |  | 10.6 (0.67)
  LS mean estimate (Brolucizumab 6 mg vs. Aflibercept 2 mg): number analyzed (Participants) | 0 | 189 | 187
  LS mean estimate (Brolucizumab 6 mg vs. Aflibercept 2 mg) |  | 9.2 (0.57) | 10.5 (0.57)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Non-Inferiority — Non-inferiority (4-letter margin); p < 0.001, ANOVA — 1-sided p-value; LS mean difference = -1.3, 95% CI 2-sided [-2.9 to 0.3], Standard Error of Mean 0.81
Statistical Analysis 2: Comparison: Brolucizumab 3 mg vs Aflibercept 2 mg; Test type: Non-Inferiority — Non-inferiority (4-letter margin); p = 0.227, ANOVA — 1-sided p-value; LS mean difference = -3.3, 95% CI 2-sided [-5.1 to -1.4], Standard Error of Mean 0.94

2. Secondary Outcome: Average Change From Baseline in BCVA Over the Period Week 40 Through Week 52
Description: BCVA will be assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts.
  Visual function of the study eye was assessed using the ETDRS protocol. Participants with a BCVA ETDRS letter score of 78 to 23 (per the inclusion criteria) (approximate Snellen equivalent of 20/32 to 20/320) in the study eye were included.
  Min and max possible scores are 0-100 respectively. A higher score represents better visual functioning.
  This endpoint was analyzed via the pairwise ANOVA method where the 2 dose groups of Brolucizumab are compared to Aflibercept.
Time Frame: Baseline and Week 40 through Week 52 (average)
Population: Full analysis set (FAS) - Observed.
  This endpoint was analyzed via the pairwise ANOVA method where the 2 dose groups of Brolucizumab are compared to Aflibercept
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 190 | 189 | 187
Scores on a scale
  LS mean estimate (Brolucizumab 3 mg vs. Aflibercept 2 mg): number analyzed (Participants) | 190 | 0 | 187
  LS mean estimate (Brolucizumab 3 mg vs. Aflibercept 2 mg) | 7.0 (0.63) |  | 10.5 (0.64)
  LS mean estimate (Brolucizumab 6 mg vs. Aflibercept 2 mg): number analyzed (Participants) | 0 | 189 | 187
  LS mean estimate (Brolucizumab 6 mg vs. Aflibercept 2 mg) |  | 9.0 (0.53) | 10.5 (0.53)
Statistical Analysis 1: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Non-Inferiority — Non-inferiority (4-letter margin); p < 0.001, ANOVA — (1-sided); Mean Difference (Net) = -1.5, 95% CI 2-sided [-3.0 to -0.0], Standard Error of Mean 0.75
Statistical Analysis 2: Comparison: Brolucizumab 3 mg vs Aflibercept 2 mg; Test type: Non-Inferiority — Non-inferiority (4-letter margin); ANOVA — (1-sided); Mean Difference (Net) = -3.5, 95% CI 2-sided [-5.2 to -1.7], Standard Error of Mean 0.90

3. Secondary Outcome: Patients Maintained at q12w - Probability of Maintaining on q12w
Description: Positive treatment status is defined as intravitreal (IVT) injections per planned dosing regimen [every 12 weeks (q12w)]. This outcome measure is pre-specified for brolucizumab treatment arms only.
Time Frame: Baseline (Week 0), Weeks 32, 36 and 48
Population: FAS - Efficacy/Safety approach
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg
Number analyzed (Participants) | 190 | 189
Probability
  Prob. of maintaining on q12w - Week 0 | 1 [NA to NA] — CIs are not applicable for probability = 1. | 1 [NA to NA] — CIs are not applicable for probability = 1.
  Prob. of maintaining on q12w - Week 32 | 0.758 [0.685 to 0.816] | 0.807 [0.739 to 0.860]
  Prob. of maintaining on q12w - Week 36 | 0.545 [0.463 to 0.619] | 0.628 [0.548 to 0.698]
  Prob. of maintaining on q12w - Week 48 | 0.474 [0.393 to 0.551] | 0.550 [0.468 to 0.625]

4. Secondary Outcome: Patients Maintained at q12w (for Those Patients Who Qualified for q12w at Week 36) - Probability of Maintaining on q12w
Description: Positive treatment status is defined as intravitreal (IVT) injections per planned dosing regimen [every 8 weeks (q8w)]. This outcome measure is pre-specified for brolucizumab treatment arms only.
Time Frame: Weeks 36 and 48
Population: FAS - Efficacy/Safety approach
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg
Number analyzed (Participants) | 190 | 189
Probability
  Prob. of maintaining on q12w - Week 36 | 1 [NA to NA] — CIs are not applicable for probability = 1. | 1 [NA to NA] — CIs are not applicable for probability = 1.
  Prob. of maintaining on q12w - Week 48 | 0.870 [0.772 to 0.928] | 0.876 [0.788 to 0.930]

5. Secondary Outcome: Change From Baseline in BCVA at Each Visit up to Week 52
Description: BCVA was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts.
  Visual function of the study eye was assessed using the ETDRS protocol. Participants with a BCVA ETDRS letter score of 78 to 23 (approximate Snellen equivalent of 20/32 to 20/320) in the study eye were included.
  Min and max possible scores are 0-100 respectively. A higher score represents better visual functioning.
Time Frame: Baseline (Week 0), Weeks 4, 6, 8, 12, 16, 18, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: Full analysis set (FAS)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 187 | 186 | 185
Scores on a scale
  Week 4 (n=187, 186, 185) | 4.0 (5.02) | 4.5 (5.22) | 5.1 (6.74)
  Week 6 (n=185,186,180): number analyzed (Participants) | 185 | 186 | 180
  Week 6 (n=185,186,180) | 5.1 (5.86) | 6.0 (6.22) | 6.8 (6.80)
  Week 8 (n=183,184,181): number analyzed (Participants) | 183 | 184 | 181
  Week 8 (n=183,184,181) | 5.6 (5.90) | 6.6 (6.54) | 7.1 (7.57)
  Week 12 (n=183,186,182): number analyzed (Participants) | 183 | 186 | 182
  Week 12 (n=183,186,182) | 6.7 (5.93) | 7.3 (6.57) | 8.1 (7.63)
  Week 16 (n=173,179,179): number analyzed (Participants) | 173 | 179 | 179
  Week 16 (n=173,179,179) | 7.0 (7.00) | 7.5 (6.83) | 8.5 (7.36)
  Week 18 (n=175,181,172): number analyzed (Participants) | 175 | 181 | 172
  Week 18 (n=175,181,172) | 7.6 (6.35) | 8.0 (6.84) | 8.8 (7.27)
  Week 20 (n=176,177,176): number analyzed (Participants) | 176 | 177 | 176
  Week 20 (n=176,177,176) | 7.8 (7.59) | 8.3 (7.51) | 9.8 (7.47)
  Week 24 (n=174,178,177): number analyzed (Participants) | 174 | 178 | 177
  Week 24 (n=174,178,177) | 8.1 (6.42) | 9.3 (7.08) | 9.2 (7.84)
  Week 28 (n=170,175,170): number analyzed (Participants) | 170 | 175 | 170
  Week 28 (n=170,175,170) | 8.2 (6.58) | 9.6 (7.40) | 10.3 (7.26)
  Week 32 (n=155,161,162): number analyzed (Participants) | 155 | 161 | 162
  Week 32 (n=155,161,162) | 8.2 (7.76) | 9.2 (7.20) | 9.9 (7.89)
  Week 36 (n=154,166,165): number analyzed (Participants) | 154 | 166 | 165
  Week 36 (n=154,166,165) | 6.9 (8.10) | 8.6 (8.15) | 10.2 (7.84)
  Week 40 (n=160,163,163): number analyzed (Participants) | 160 | 163 | 163
  Week 40 (n=160,163,163) | 7.3 (10.47) | 9.5 (7.99) | 10.0 (8.28)
  Week 44 (n=156,157,163): number analyzed (Participants) | 156 | 157 | 163
  Week 44 (n=156,157,163) | 7.5 (10.92) | 9.6 (7.66) | 10.7 (8.25)
  Week 48 (n=155,154,159): number analyzed (Participants) | 155 | 154 | 159
  Week 48 (n=155,154,159) | 7.2 (11.53) | 10.0 (7.63) | 11.1 (8.75)
  Week 52 (n=156,153,160): number analyzed (Participants) | 156 | 153 | 160
  Week 52 (n=156,153,160) | 7.8 (10.72) | 10.2 (7.66) | 10.7 (8.87)

6. Secondary Outcome: BCVA (Letters Read): ANOVA Results for Average Change From Baseline Over the Period Week 88 Through Week 100 for the Study Eye (FAS - LOCF)
Description: Visual acuity was assessed at every study visit using best correction determined from protocol refraction (BCVA). BCVA measurements were taken in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity testing charts.
  LS Mean estimates are reported, comparing the 2 Brolucizumab arms to Aflibercept. Results do not apply to the Brolucizumab 6 mg arm when Brolucizumab 3mg is compared to Aflibercept. Likewise, results do not apply to the Brolucizumab 3 mg arm when Brolucizumab 6 mg is compared to Aflibercept.
Time Frame: Baseline, and Week 88 through Week 100 (average)
Population: Full Analysis Set - LOCF
Measure: Least Squares Mean (Standard Error); unit: BCVA letters read
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 190 | 189 | 187
BCVA letters read
  LS mean estimate (Brolucizumab 3 mg vs Aflibercept 2 mg) (n=190, 0, 187): number analyzed (Participants) | 190 | 0 | 187
  LS mean estimate (Brolucizumab 3 mg vs Aflibercept 2 mg) (n=190, 0, 187) | 6.7 (0.77) |  | 10.6 (0.78)
  LS mean estimate (Brolucizumab 6 mg vs Aflibercept 2 mg) (n=0, 189,187): number analyzed (Participants) | 0 | 189 | 187
  LS mean estimate (Brolucizumab 6 mg vs Aflibercept 2 mg) (n=0, 189,187) |  | 8.6 (0.72) | 10.6 (0.73)
Statistical Analysis 1: Comparison: Brolucizumab 3 mg vs Aflibercept 2 mg; Test type: Other — Descriptive; ANOVA; LS mean difference = -3.8, 95% CI 2-sided [-6.0 to -1.7], Standard Error of Mean 1.09
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Other — Descriptive; ANOVA; LS mean difference = -2.0, 95% CI 2-sided [-4.0 to 0.1], Standard Error of Mean 1.03

7. Secondary Outcome: Patients Maintained at q12w up to Week 64 (After Three q12w- Treatment Intervals) and Week 100 - Probability of Maintaining on q12w
Description: This outcome measure is pre-specified for brolucizumab treatment arms only
Time Frame: Baseline (Week 0), Weeks 32, 36, 48, 60, 72, 84, and 96
Population: FAS - Efficacy/Safety approach
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 190 | 189 | 0
Probability
  Prob. of maintaining on q12w - Week 0 | 1 [NA to NA] — Not applicable when probability = 1 | 1 [NA to NA] — Not applicable when probability = 1 |
  Prob. of maintaining on q12w - Week 32 | 0.758 [0.685 to 0.816] | 0.807 [0.739 to 0.860] |
  Prob. of maintaining on q12w - Week 36 | 0.545 [0.463 to 0.619] | 0.628 [0.548 to 0.698] |
  Prob. of maintaining on q12w - Week 48 | 0.474 [0.393 to 0.551] | 0.550 [0.468 to 0.625] |
  Prob. of maintaining on q12w - Week 60 | 0.403 [0.323 to 0.482] | 0.520 [0.437 to 0.596] |
  Prob. of maintaining on q12w - Week 72 | 0.394 [0.314 to 0.473] | 0.487 [0.404 to 0.565] |
  Prob. of maintaining on q12w - Week 84 | 0.365 [0.285 to 0.445] | 0.460 [0.376 to 0.539] |
  Prob. of maintaining on q12w - Week 96 | 0.334 [0.254 to 0.415] | 0.441 [0.357 to 0.521] |

8. Secondary Outcome: Secondary: Patients Maintained at q12w up to Week 64 (After Three q12w- Treatment Intervals) and Week 100, Within Those Patients That Qualified for q12w at Week 36 - Probability of Maintaining on q12w
Description: This outcome measure is pre-specified for brolucizumab treatment arms only
Time Frame: Baseline (Week 0), Weeks 32, 36, 48, 60, 72, 84, and 96
Population: FAS - Efficacy/Safety approach
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 190 | 189 | 0
Probability
  Prob. of maintaining on q12w - Week 0 | 1 [NA to NA] — Not applicable when probability = 1 | 1 [NA to NA] — Not applicable when probability = 1 |
  Prob. of maintaining on q12w - Week 32 | 1 [NA to NA] — Not applicable when probability = 1 | 1 [NA to NA] — Not applicable when probability = 1 |
  Prob. of maintaining on q12w - Week 36 | 1 [NA to NA] — Not applicable when probability = 1 | 1 [NA to NA] — Not applicable when probability = 1 |
  Prob. of maintaining on q12w - Week 48 | 0.870 [0.772 to 0.928] | 0.876 [0.788 to 0.930] |
  Prob. of maintaining on q12w - Week 60 | 0.740 [0.622 to 0.826] | 0.828 [0.730 to 0.892] |
  Prob. of maintaining on q12w - Week 72 | 0.723 [0.603 to 0.812] | 0.775 [0.670 to 0.851] |
  Prob. of maintaining on q12w - Week 84 | 0.670 [0.544 to 0.769] | 0.732 [0.621 to 0.816] |
  Prob. of maintaining on q12w - Week 96 | 0.613 [0.482 to 0.720] | 0.702 [0.587 to 0.791] |

9. Secondary Outcome: Change From Baseline in Central Subfield Thickness (CSFT) at Each Visit up to Week 52 - Pairwise ANOVA Results
Description: Central Subfield Thickness Assessed by Spectral domain optical coherence tomography (SD-OCT) from the central reading center.
  LS Mean estimates are reported, comparing the 2 Brolucizumab arms to Aflibercept. Results do not apply to the Brolucizumab 6 mg arm when Brolucizumab 3mg is compared to Aflibercept. Likewise, results do not apply to the Brolucizumab 3 mg arm when Brolucizumab 6 mg is compared to Aflibercept.
Time Frame: Baseline up to week 52
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: μm
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 190 | 189 | 187
μm
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 4 (n=190, 0, 187): number analyzed (Participants) | 190 | 0 | 187
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 4 (n=190, 0, 187) | -104.7 (6.11) |  | -104.1 (6.15)
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg) - Week 4 (n=0, 189, 187): number analyzed (Participants) | 0 | 189 | 187
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg) - Week 4 (n=0, 189, 187) |  | -105.6 (5.92) | -103.4 (5.95)
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 6 (n=190, 0, 187): number analyzed (Participants) | 190 | 0 | 187
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 6 (n=190, 0, 187) | -107.1 (6.24) |  | -119.3 (6.29)
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg) - Week 6 (n=0, 189, 187): number analyzed (Participants) | 0 | 189 | 187
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg) - Week 6 (n=0, 189, 187) |  | -116.1 (5.89) | -118.6 (5.92)
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 8 (n=190, 0, 187): number analyzed (Participants) | 190 | 0 | 187
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 8 (n=190, 0, 187) | -125.1 (6.06) |  | -126.1 (6.11)
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg)- Week 8 (n=0, 189, 187): number analyzed (Participants) | 0 | 189 | 187
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg)- Week 8 (n=0, 189, 187) |  | -128.9 (5.82) | -125.6 (5.86)
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 12 (n=190, 0, 187): number analyzed (Participants) | 190 | 0 | 187
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 12 (n=190, 0, 187) | -131.0 (6.14) |  | -137.4 (6.19)
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg) - Week 12 (n=0, 189, 187): number analyzed (Participants) | 0 | 189 | 187
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg) - Week 12 (n=0, 189, 187) |  | -134.5 (6.22) | -137.3 (6.26)
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 16 (n=190, 0, 187): number analyzed (Participants) | 190 | 0 | 187
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 16 (n=190, 0, 187) | -142.3 (5.98) |  | -143.3 (6.02)
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg) - Week 16 (n=0, 189, 187): number analyzed (Participants) | 0 | 189 | 187
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg) - Week 16 (n=0, 189, 187) |  | -146.5 (5.83) | -143.1 (5.86)
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 18 (n=190, 0, 187): number analyzed (Participants) | 190 | 0 | 187
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 18 (n=190, 0, 187) | -138.1 (6.27) |  | -147.0 (6.32)
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg) - Week 18 (n=0, 189, 187): number analyzed (Participants) | 0 | 189 | 187
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg) - Week 18 (n=0, 189, 187) |  | -144.2 (5.96) | -146.8 (5.99)
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 20 (n=190, 0, 187): number analyzed (Participants) | 190 | 0 | 187
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 20 (n=190, 0, 187) | -151.8 (6.01) |  | -148.3 (6.06)
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg) - Week 20 (n=0, 189, 187): number analyzed (Participants) | 0 | 189 | 187
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg) - Week 20 (n=0, 189, 187) |  | -153.8 (5.71) | -148.0 (5.74)
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 24 (n=190, 0, 187): number analyzed (Participants) | 190 | 0 | 187
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 24 (n=190, 0, 187) | -152.6 (6.37) |  | -138.7 (6.42)
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg) - Week 24 (n=0, 189, 187): number analyzed (Participants) | 0 | 189 | 187
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg) - Week 24 (n=0, 189, 187) |  | -156.2 (6.30) | -138.4 (6.33)
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 28 (n=190, 0, 187): number analyzed (Participants) | 190 | 0 | 187
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 28 (n=190, 0, 187) | -163.4 (5.81) |  | -154.6 (5.85)
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg) - Week 28 (n=0, 189, 187): number analyzed (Participants) | 0 | 189 | 187
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg) - Week 28 (n=0, 189, 187) |  | -163.3 (5.97) | -154.6 (6.00)
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 32 (n=190, 0, 187): number analyzed (Participants) | 190 | 0 | 187
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 32 (n=190, 0, 187) | -147.4 (6.68) |  | -144.3 (6.73)
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg) - Week 32 (n=0, 189, 187): number analyzed (Participants) | 0 | 189 | 187
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg) - Week 32 (n=0, 189, 187) |  | -156.0 (6.35) | -144.2 (6.38)
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 36 (n=190, 0, 187): number analyzed (Participants) | 190 | 0 | 187
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 36 (n=190, 0, 187) | -119.8 (7.74) |  | -156.0 (7.81)
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg) - Week 36 (n=0, 189, 187): number analyzed (Participants) | 0 | 189 | 187
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg) - Week 36 (n=0, 189, 187) |  | -135.1 (7.01) | -155.5 (7.05)
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 40 (n=190, 0, 187): number analyzed (Participants) | 190 | 0 | 187
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 40 (n=190, 0, 187) | -155.8 (6.46) |  | -149.7 (6.51)
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg) - Week 40 (n=0, 189, 187): number analyzed (Participants) | 0 | 189 | 187
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg) - Week 40 (n=0, 189, 187) |  | -156.9 (6.68) | -150.4 (6.72)
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 44 (n=190, 0, 187): number analyzed (Participants) | 190 | 0 | 187
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 44 (n=190, 0, 187) | -155.4 (6.56) |  | -163.4 (6.62)
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg) - Week 44 (n=0, 189, 187): number analyzed (Participants) | 0 | 189 | 187
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg) - Week 44 (n=0, 189, 187) |  | -162.2 (6.17) | -163.3 (6.21)
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 48 (n=190, 0, 187): number analyzed (Participants) | 190 | 0 | 187
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 48 (n=190, 0, 187) | -144.2 (6.92) |  | -157.8 (6.98)
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg) - Week 48 (n=0, 189, 187): number analyzed (Participants) | 0 | 189 | 187
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg) - Week 48 (n=0, 189, 187) |  | -153.5 (6.52) | -158.2 (6.55)
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 52 (n=190, 0, 187): number analyzed (Participants) | 190 | 0 | 187
  LS mean estimate (Brolucizumab 3mg vs Aflibercept 2mg) - Week 52 (n=190, 0, 187) | -156.4 (6.70) |  | -160.7 (6.75)
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg) - Week 52 (n=0, 189, 187): number analyzed (Participants) | 0 | 189 | 187
  LS mean estimate (Brolucizumab 6mg vs Aflibercept 2mg) - Week 52 (n=0, 189, 187) |  | -165.5 (6.17) | -160.4 (6.21)
Statistical Analysis 1: Comparison: Brolucizumab 3 mg vs Aflibercept 2 mg; Week 4; Test type: Other — Descriptive; ANOVA; LS mean difference = -0.7, 95% CI 2-sided [-17.7 to 16.4], Standard Error of Mean 8.68
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 4; Test type: Other — Descriptive; ANOVA; LS mean difference = -2.1, 95% CI 2-sided [-18.7 to 14.4], Standard Error of Mean 8.41
Statistical Analysis 3: Comparison: Brolucizumab 3 mg vs Aflibercept 2 mg; Week 6; Test type: Other — Descriptive; ANOVA; LS mean difference = 12.2, 95% CI 2-sided [-5.2 to 29.7], Standard Error of Mean 8.87
Statistical Analysis 4: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 6; Test type: Other — Descriptive; ANOVA; LS mean difference = 2.4, 95% CI 2-sided [-14.0 to 18.9], Standard Error of Mean 8.38
Statistical Analysis 5: Comparison: Brolucizumab 3 mg vs Aflibercept 2 mg; Week 8; Test type: Other — Descriptive; ANOVA; LS mean difference = 1.0, 95% CI 2-sided [-16.0 to 17.9], Standard Error of Mean 8.61
Statistical Analysis 6: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 8; Test type: Other — Descriptive; ANOVA; LS mean difference = -3.4, 95% CI 2-sided [-19.6 to 12.9], Standard Error of Mean 8.28
Statistical Analysis 7: Comparison: Brolucizumab 3 mg vs Aflibercept 2 mg; Week 12; Test type: Other — Descriptive; ANOVA; LS mean difference = 6.4, 95% CI 2-sided [-10.7 to 23.6], Standard Error of Mean 8.73
Statistical Analysis 8: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 12; Test type: Other — Descriptive; ANOVA; LS mean difference = 2.8, 95% CI 2-sided [-14.6 to 20.2], Standard Error of Mean 8.85
Statistical Analysis 9: Comparison: Brolucizumab 3 mg vs Aflibercept 2 mg; Week 16; Test type: Other — Descriptive; ANOVA; LS mean difference = 1.0, 95% CI 2-sided [-15.7 to 17.8], Standard Error of Mean 8.50
Statistical Analysis 10: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 16; Test type: Other — Descriptive; ANOVA; LS mean difference = -3.4, 95% CI 2-sided [-19.7 to 12.9], Standard Error of Mean 8.29
Statistical Analysis 11: Comparison: Brolucizumab 3 mg vs Aflibercept 2 mg; Week 18; Test type: Other — Descriptive; ANOVA; LS mean difference = 8.9, 95% CI 2-sided [-8.6 to 26.5], Standard Error of Mean 8.92
Statistical Analysis 12: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 18; Test type: Other — Descriptive; ANOVA; LS mean difference = 2.6, 95% CI 2-sided [-14.1 to 19.2], Standard Error of Mean 8.47
Statistical Analysis 13: Comparison: Brolucizumab 3 mg vs Aflibercept 2 mg; Week 20; Test type: Other — Descriptive; ANOVA; LS mean difference = -3.4, 95% CI 2-sided [-20.2 to 13.4], Standard Error of Mean 8.55
Statistical Analysis 14: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 20; Test type: Other — Descriptive; ANOVA; LS mean difference = -5.8, 95% CI 2-sided [-21.7 to 10.2], Standard Error of Mean 8.12
Statistical Analysis 15: Comparison: Brolucizumab 3 mg vs Aflibercept 2 mg; Week 24; Test type: Other — Descriptive; ANOVA; LS mean difference = -13.9, 95% CI 2-sided [-31.7 to 3.9], Standard Error of Mean 9.06
Statistical Analysis 16: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 24; Test type: Other — Descriptive; ANOVA; LS mean difference = -17.8, 95% CI 2-sided [-35.4 to -0.2], Standard Error of Mean 8.95
Statistical Analysis 17: Comparison: Brolucizumab 3 mg vs Aflibercept 2 mg; Week 28; Test type: Other — Descriptive; ANOVA; LS mean difference = -8.7, 95% CI 2-sided [-25.0 to 7.5], Standard Error of Mean 8.26
Statistical Analysis 18: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 28; Test type: Other — Descriptive; ANOVA; LS mean difference = -8.7, 95% CI 2-sided [-25.4 to 8.0], Standard Error of Mean 8.49
Statistical Analysis 19: Comparison: Brolucizumab 3 mg vs Aflibercept 2 mg; Week 32; Test type: Other — Descriptive; ANOVA; LS mean difference = -3.2, 95% CI 2-sided [-21.8 to 15.5], Standard Error of Mean 9.49
Statistical Analysis 20: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 32; Test type: Other — Descriptive; ANOVA; LS mean difference = -11.7, 95% CI 2-sided [-29.5 to 6.0], Standard Error of Mean 9.02
Statistical Analysis 21: Comparison: Brolucizumab 3 mg vs Aflibercept 2 mg; Week 36; Test type: Other — Descriptive; ANOVA; LS mean difference = 36.3, 95% CI 2-sided [14.6 to 57.9], Standard Error of Mean 11.01
Statistical Analysis 22: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 36; Test type: Other — Descriptive; ANOVA; LS mean difference = 20.4, 95% CI 2-sided [0.7 to 40.0], Standard Error of Mean 9.97
Statistical Analysis 23: Comparison: Brolucizumab 3 mg vs Aflibercept 2 mg; Week 40; Test type: Other — Descriptive; ANOVA; LS mean difference = -6.1, 95% CI 2-sided [-24.2 to 11.9], Standard Error of Mean 9.19
Statistical Analysis 24: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 40; Test type: Other — Descriptive; ANOVA; LS mean difference = -6.5, 95% CI 2-sided [-25.2 to 12.2], Standard Error of Mean 9.50
Statistical Analysis 25: Comparison: Brolucizumab 3 mg vs Aflibercept 2 mg; Week 44; Test type: Other — Descriptive; ANOVA; LS mean difference = 7.9, 95% CI 2-sided [-10.4 to 26.3], Standard Error of Mean 9.33
Statistical Analysis 26: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 44; Test type: Other — Descriptive; ANOVA; LS mean difference = 1.1, 95% CI 2-sided [-16.2 to 18.3], Standard Error of Mean 8.78
Statistical Analysis 27: Comparison: Brolucizumab 3 mg vs Aflibercept 2 mg; Week 48; Test type: Other — Descriptive; ANOVA; LS mean difference = 13.6, 95% CI 2-sided [-5.8 to 32.9], Standard Error of Mean 9.84
Statistical Analysis 28: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 48; Test type: Other — Descriptive; ANOVA; LS mean difference = 4.7, 95% CI 2-sided [-13.5 to 23.0], Standard Error of Mean 9.26
Statistical Analysis 29: Comparison: Brolucizumab 3 mg vs Aflibercept 2 mg; Week 52; Test type: Other — Descriptive; ANOVA; LS mean difference = 4.3, 95% CI 2-sided [-14.5 to 23.0], Standard Error of Mean 9.52
Statistical Analysis 30: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Week 52; Test type: Other — Descriptive; ANOVA; LS mean difference = -5.1, 95% CI 2-sided [-22.3 to 12.2], Standard Error of Mean 8.78

10. Secondary Outcome: Central Subfield Thickness (CSFT) (Micrometers): ANOVA Results for Average Change From Baseline Over the Period Week 88 Through Week 100 for the Study Eye (Full Analysis Set - LOCF)
Description: Central subfield thickness (average thickness of circular 1mm area centered around fovea measured from RPE to ILM, inclusively). Assessed with Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts.
  LS Mean estimates are reported, comparing the 2 Brolucizumab arms to Aflibercept. Results do not apply to the Brolucizumab 6 mg arm when Brolucizumab 3mg is compared to Aflibercept. Likewise, results do not apply to the Brolucizumab 3 mg arm when Brolucizumab 6 mg is compared to Aflibercept.
Time Frame: Baseline, and Week 88 through Week 100 (average)
Population: Full Analysis Set - LOCF
Measure: Least Squares Mean (Standard Error); unit: micrometers
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 190 | 189 | 187
micrometers
  LS mean estimate (Brolucizumab 3 mg vs Aflibercept 2 mg) (n=190, 0, 187): number analyzed (Participants) | 190 | 0 | 187
  LS mean estimate (Brolucizumab 3 mg vs Aflibercept 2 mg) (n=190, 0, 187) | -167.1 (6.54) |  | -168.8 (6.59)
  LS mean estimate (Brolucizumab 6 mg vs Aflibercept 2 mg) (n=0, 189,187): number analyzed (Participants) | 0 | 189 | 187
  LS mean estimate (Brolucizumab 6 mg vs Aflibercept 2 mg) (n=0, 189,187) |  | -171.9 (6.18) | -168.5 (6.22)
Statistical Analysis 1: Comparison: Brolucizumab 3 mg vs Aflibercept 2 mg; Test type: Other — Descriptive; ANOVA; LS mean difference = 1.7, 95% CI 2-sided [-16.6 to 20.0], Standard Error of Mean 9.30
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Other — Descriptive; ANOVA; LS mean difference = -3.5, 95% CI 2-sided [-20.7 to 13.8], Standard Error of Mean 8.79

11. Secondary Outcome: Number of Patients With Presence of Subretinal Fluid (SRF) at Each Assessment Visit
Description: Subretinal Fluid (SRF) status in the central subfield: proportion of subjects with presence of SRF in the study eye by visit
Time Frame: Baseline up to Week 52 and Week 100
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 190 | 189 | 187
Participants
  Week 4 | 26 | 23 | 27
  Week 6 | 20 | 17 | 17
  Week 8 | 10 | 9 | 12
  Week 12 | 11 | 8 | 8
  Week16 | 6 | 6 | 7
  Week18 | 7 | 4 | 6
  Week 20 | 5 | 4 | 6
  Week 24 | 7 | 3 | 6
  Week 28 | 5 | 2 | 3
  Week 32 | 11 | 1 | 6
  Week 36 | 16 | 14 | 4
  Week 40 | 8 | 5 | 6
  Week 44 | 4 | 4 | 4
  Week 48 | 7 | 8 | 3
  Week 52 | 4 | 4 | 4
  Week 56 | 9 | 3 | 5
  Week 60 | 9 | 5 | 5
  Week 64 | 6 | 4 | 5
  Week 68 | 6 | 4 | 3
  Week 72 | 5 | 4 | 4
  Week 76 | 4 | 4 | 4
  Week 80 | 5 | 4 | 5
  Week 84 | 6 | 3 | 3
  Week 88 | 7 | 2 | 4
  Week 92 | 4 | 2 | 4
  Week 96 | 5 | 3 | 5
  Week 100 | 3 | 2 | 2

12. Secondary Outcome: Number of Patients With Presence of Intraretinal Fluid (IRF) at Each Assessment Visit
Description: Intraretinal Fluid (IRF) status in the central subfield: proportion of subjects with presence of IRF in the study eye by visit
Time Frame: Baseline, up to Week 52 and Week 100
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 190 | 189 | 187
Participants
  Week 4 | 176 | 169 | 169
  Week 6 | 177 | 169 | 169
  Week 8 | 166 | 161 | 164
  Week 12 | 167 | 162 | 165
  Week 16 | 155 | 150 | 156
  Week 18 | 152 | 149 | 154
  Week 20 | 142 | 147 | 145
  Week 24 | 142 | 140 | 153
  Week 28 | 139 | 130 | 144
  Week 32 | 143 | 131 | 156
  Week 36 | 153 | 141 | 144
  Week 40 | 129 | 114 | 150
  Week 44 | 127 | 118 | 135
  Week 48 | 132 | 123 | 147
  Week 52 | 113 | 114 | 137
  Week 56 | 111 | 103 | 138
  Week 60 | 119 | 115 | 126
  Week 64 | 102 | 105 | 131
  Week 68 | 109 | 98 | 118
  Week 72 | 107 | 103 | 126
  Week 76 | 98 | 96 | 118
  Week 80 | 96 | 85 | 120
  Week 84 | 102 | 92 | 108
  Week 88 | 89 | 85 | 114
  Week 92 | 91 | 86 | 105
  Week 96 | 92 | 90 | 107
  Week 100 | 87 | 79 | 101

13. Secondary Outcome: Number of Patients With Presence of SRF and/or IRF in the Study Eye by Visit
Description: Subretinal Fluid (SRF) and Intraretinal Fluid (IRF) status in the central subfield: proportion of subjects with presence of SRF and/or IRF in the study eye by visit
Time Frame: Baseline, up to Week 52 and Week 100
Population: Full analysis set (FAS) - Last observation carried forward (LOCF)
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 190 | 189 | 187
Participants
  Week 4 | 177 | 172 | 171
  Week 6 | 177 | 173 | 169
  Week 8 | 166 | 162 | 164
  Week 12 | 168 | 162 | 165
  Week 16 | 156 | 150 | 156
  Week 18 | 153 | 149 | 154
  Week 20 | 142 | 147 | 145
  Week 24 | 142 | 140 | 153
  Week 28 | 139 | 130 | 144
  Week 32 | 143 | 131 | 156
  Week 36 | 153 | 141 | 144
  Week 40 | 129 | 114 | 150
  Week 44 | 127 | 118 | 135
  Week 48 | 132 | 123 | 147
  Week 52 | 113 | 114 | 137
  Week 56 | 111 | 103 | 138
  Week 60 | 120 | 115 | 126
  Week 64 | 102 | 105 | 131
  Week 68 | 109 | 98 | 118
  Week 72 | 107 | 103 | 126
  Week 76 | 98 | 96 | 118
  Week 80 | 96 | 85 | 120
  Week 84 | 102 | 92 | 108
  Week 88 | 89 | 85 | 114
  Week 92 | 91 | 86 | 105
  Week 96 | 92 | 90 | 107
  Week 100 | 87 | 79 | 101

14. Secondary Outcome: Number of Patients With Presence of Leakage on Fluorescein Angiography (FA) at Week 52
Description: Assessed by angiography.
Time Frame: Week 52
Population: Full analysis set (FAS) - Last observation carried forward (LOCF). The angiogram results are not available at baseline on all participants because in rare cases, the images could not be read e.g., because of poor quality.
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 189 | 188 | 186
Participants | 114 | 108 | 140

15. Secondary Outcome: Number of Patients With Presence of Leakage on Fluorescein Angiography (FA) at Week 100
Description: Assessed by angiography.
Time Frame: Week 100
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 190 | 188 | 186
Participants | 94 | 80 | 104

16. Secondary Outcome: Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS): Number of Subjects With >=2-step Improvement From Baseline in the DRSS Score at Each Assessment Visit for the Study Eye - Number of Subjects
Description: Severity of Diabetic Retinopathy (DR) was evaluated using the ETDRS DRSS score assessed by the Central Reading Center (CRC) based on color fundus photography images in the study eye. When the ETDRS-DR severities were evaluable, they were categorized on a 12-level scale, from 1 (DR absent) to 12 (very advanced PDR). A lower score represents better visual functioning.
Time Frame: Baseline, Weeks 28, 52, 76, 100
Population: Full analysis set (FAS) - Last observation carried forward (LOCF). The results are not available at baseline on all participants because in rare cases, the images could not be read e.g., because of poor quality.
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 185 | 186 | 184
Participants
  Week 28 | 44 | 49 | 39
  Week 52 | 53 | 55 | 40
  Week 76 | 59 | 55 | 51
  Week 100 | 60 | 61 | 54

17. Secondary Outcome: Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS): Proportion of Subjects With >=2-step Improvement From Baseline in the DRSS Score at Each Assessment Visit for the Study Eye - Percentage Estimates
Description: Severity of Diabetic Retinopathy (DR) was evaluated using the ETDRS DRSS score assessed by the Central Reading Center (CRC) based on color fundus photography images in the study eye. When the ETDRS-DR severities were evaluable, they were categorized on a 12-level scale, from 1 (DR absent) to 12 (very advanced PDR). A lower score represents better visual functioning.
  * estimates are reported, comparing the 2 Brolucizumab arms to Aflibercept. Results do not apply to the Brolucizumab 6 mg arm when Brolucizumab 3mg is compared to Aflibercept. Likewise, results do not apply to the Brolucizumab 3 mg arm when Brolucizumab 6 mg is compared to Aflibercept.
  * estimates represent the % of participants who were estimated to have a ">=2-step Improvement From Baseline in the DRSS Score" from pairwise logistic regression models adjusting for baseline DRSS score categories (<=4, ≥5), age categories (<65, ≥65 years) and treatment as fixed effect factors.
  Abbreviation: Proportion Estimates = P.E.
Time Frame: Baseline, Weeks 28, 52, 76, 100
Population: as for outcome 16
Measure: Number; unit: Percentage estimates
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 185 | 186 | 184
Percentage estimates
  Comparison of Brolucizumab 3 mg vs. Aflibercept 2 mg - P.E. (%) at Week 28 (n = 185,0, 184): number analyzed (Participants) | 185 | 0 | 184
  Comparison of Brolucizumab 3 mg vs. Aflibercept 2 mg - P.E. (%) at Week 28 (n = 185,0, 184) | 23.3 |  | 21.7
  Comparison of Brolucizumab 6 mg vs. Aflibercept 2 mg - P.E.(%) at Week 28 (n = 0, 186, 184): number analyzed (Participants) | 0 | 186 | 184
  Comparison of Brolucizumab 6 mg vs. Aflibercept 2 mg - P.E.(%) at Week 28 (n = 0, 186, 184) |  | 25.8 | 21.7
  Comparison of Brolucizumab 3 mg vs. Aflibercept 2 mg - P.E. (%) at Week 52 (n = 185,0, 184): number analyzed (Participants) | 185 | 0 | 184
  Comparison of Brolucizumab 3 mg vs. Aflibercept 2 mg - P.E. (%) at Week 52 (n = 185,0, 184) | 28.0 |  | 22.3
  Comparison of Brolucizumab 6 mg vs. Aflibercept 2 mg - P.E. (%) at Week 52 (n = 0, 186, 184): number analyzed (Participants) | 0 | 186 | 184
  Comparison of Brolucizumab 6 mg vs. Aflibercept 2 mg - P.E. (%) at Week 52 (n = 0, 186, 184) |  | 29.0 | 22.2
  Comparison of Brolucizumab 3 mg vs. Aflibercept 2 mg - P.E. (%) at Week 76 (n = 185,0, 184): number analyzed (Participants) | 185 | 0 | 184
  Comparison of Brolucizumab 3 mg vs. Aflibercept 2 mg - P.E. (%) at Week 76 (n = 185,0, 184) | 31.2 |  | 28.4
  Comparison of Brolucizumab 6 mg vs. Aflibercept 2 mg - P.E.(%) at Week 76 (n = 0, 186, 184): number analyzed (Participants) | 0 | 186 | 184
  Comparison of Brolucizumab 6 mg vs. Aflibercept 2 mg - P.E.(%) at Week 76 (n = 0, 186, 184) |  | 29.0 | 28.3
  Comparison of Brolucizumab 3 mg vs. Aflibercept 2 mg - P.E. (%) at Week 100 (n = 185,0, 184): number analyzed (Participants) | 185 | 0 | 184
  Comparison of Brolucizumab 3 mg vs. Aflibercept 2 mg - P.E. (%) at Week 100 (n = 185,0, 184) | 31.7 |  | 30.1
  Comparison of Brolucizumab 6 mg vs. Aflibercept 2 mg - P.E.(%) at Week 100 (n = 0, 186, 184): number analyzed (Participants) | 0 | 186 | 184
  Comparison of Brolucizumab 6 mg vs. Aflibercept 2 mg - P.E.(%) at Week 100 (n = 0, 186, 184) |  | 32.1 | 30.0
Statistical Analysis 1: Comparison: Brolucizumab 3 mg vs Aflibercept 2 mg; Test type: Other — Descriptive; Week 28; Bootstrap method; Difference - % = 1.6, 95% CI 2-sided [-5.3 to 8.4]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Other — Descriptive; Week 28; Bootstrap method; Difference - % = 4.1, 95% CI 2-sided [-2.1 to 10.3]
Statistical Analysis 3: Comparison: Brolucizumab 3 mg vs Aflibercept 2 mg; Test type: Other — Descriptive; Week 52; Bootstrap method; Difference - % = 5.8, 95% CI 2-sided [-1.2 to 12.4]
Statistical Analysis 4: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Other — Descriptive; Week 52; Bootstrap method; Difference - % = 6.7, 95% CI 2-sided [0.6 to 12.9]
Statistical Analysis 5: Comparison: Brolucizumab 3 mg vs Aflibercept 2 mg; Test type: Other — Descriptive: Week 76; Bootstrap method; Difference - % = 2.8, 95% CI 2-sided [-3.9 to 9.4]
Statistical Analysis 6: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Other — Descriptive: Week 76; Bootstrap method; Difference - % = 0.7, 95% CI 2-sided [-5.7 to 7.0]
Statistical Analysis 7: Comparison: Brolucizumab 3 mg vs Aflibercept 2 mg; Test type: Other — Descriptive: Week 100; Bootstrap method; Difference - % = 1.7, 95% CI 2-sided [-5.0 to 8.1]
Statistical Analysis 8: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Other — Descriptive: Week 100; Bootstrap method; Difference - % = 2.2, 95% CI 2-sided [-4.0 to 8.4]

18. Secondary Outcome: Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS): Number of Subjects With >=3-step Improvement From Baseline in the DRSS Score at Each Assessment Visit for the Study Eye - Number of Subjects
Description: as for outcome 16
Time Frame: Baseline, Weeks 28, 52, 76, 100
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 185 | 186 | 184
Participants
  Week 28 | 23 | 32 | 22
  Week 52 | 24 | 39 | 30
  Week 76 | 27 | 40 | 42
  Week 100 | 29 | 44 | 41

19. Secondary Outcome: Early Treatment Diabetic Retinopathy Study (ETDRS) Diabetic Retinopathy Severity Scale (DRSS): Proportion of Subjects With >=3-step Improvement From Baseline in the DRSS Score at Each Assessment Visit for the Study Eye - Percentage Estimates
Description: Severity of Diabetic Retinopathy (DR) was evaluated using the ETDRS DRSS score assessed by the Central Reading Center (CRC) based on color fundus photography images in the study eye. When the ETDRS-DR severities were evaluable, they were categorized on a 12-level scale, from 1 (DR absent) to 12 (very advanced PDR). A lower score represents better visual functioning.
  * estimates are reported, comparing the 2 Brolucizumab arms to Aflibercept. Results do not apply to the Brolucizumab 6 mg arm when Brolucizumab 3mg is compared to Aflibercept. Likewise, results do not apply to the Brolucizumab 3 mg arm when Brolucizumab 6 mg is compared to Aflibercept.
  * estimates represent the % of participants who were estimated to have a ">=3-step Improvement From Baseline in the DRSS Score" from pairwise logistic regression models adjusting for baseline DRSS score categories (<=4, ≥5), age categories (<65, ≥65 years) and treatment as fixed effect factors.
  Abbreviation: Proportion Estimates = P.E.
Time Frame: Baseline, Weeks 28, 52, 76, 100
Population: as for outcome 16
Measure: Number; unit: Percentage estimates
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 185 | 186 | 184
Percentage estimates
  Comparison of Brolucizumab 3 mg vs. Aflibercept 2 mg - P.E. (%) at Week 28 (n = 185, 0, 184): number analyzed (Participants) | 185 | 0 | 184
  Comparison of Brolucizumab 3 mg vs. Aflibercept 2 mg - P.E. (%) at Week 28 (n = 185, 0, 184) | 12.1 |  | 12.3
  Comparison of Brolucizumab 6 mg vs. Aflibercept 2 mg - P.E. (%) at Week 28 (n = 0, 186, 184): number analyzed (Participants) | 0 | 186 | 184
  Comparison of Brolucizumab 6 mg vs. Aflibercept 2 mg - P.E. (%) at Week 28 (n = 0, 186, 184) |  | 16.8 | 12.2
  Comparison of Brolucizumab 3 mg vs. Aflibercept 2 mg - P.E.(%) at Week 52 (n = 185, 0, 184): number analyzed (Participants) | 185 | 0 | 184
  Comparison of Brolucizumab 3 mg vs. Aflibercept 2 mg - P.E.(%) at Week 52 (n = 185, 0, 184) | 12.6 |  | 16.8
  Comparison of Brolucizumab 6 mg vs. Aflibercept 2 mg - P.E. (%) at Week 52 (n = 0, 186, 184): number analyzed (Participants) | 0 | 186 | 184
  Comparison of Brolucizumab 6 mg vs. Aflibercept 2 mg - P.E. (%) at Week 52 (n = 0, 186, 184) |  | 20.5 | 16.7
  Comparison of Brolucizumab 3 mg vs. Aflibercept 2 mg - P.E. (%) at Week 76 (n = 185, 0, 184): number analyzed (Participants) | 185 | 0 | 184
  Comparison of Brolucizumab 3 mg vs. Aflibercept 2 mg - P.E. (%) at Week 76 (n = 185, 0, 184) | 14.2 |  | 23.4
  Comparison of Brolucizumab 6 mg vs. Aflibercept 2 mg - P.E. (%) at Week 76 (n = 0, 186, 184): number analyzed (Participants) | 0 | 186 | 184
  Comparison of Brolucizumab 6 mg vs. Aflibercept 2 mg - P.E. (%) at Week 76 (n = 0, 186, 184) |  | 21.1 | 23.3
  Comparison of Brolucizumab 3 mg vs. Aflibercept 2 mg - P.E. (%) at Week 100 (n = 185, 0, 184): number analyzed (Participants) | 185 | 0 | 184
  Comparison of Brolucizumab 3 mg vs. Aflibercept 2 mg - P.E. (%) at Week 100 (n = 185, 0, 184) | 15.2 |  | 22.9
  Comparison of Brolucizumab 6 mg vs. Aflibercept 2 mg - P.E. (%) at Week 100 (n = 0, 186, 184): number analyzed (Participants) | 0 | 186 | 184
  Comparison of Brolucizumab 6 mg vs. Aflibercept 2 mg - P.E. (%) at Week 100 (n = 0, 186, 184) |  | 23.2 | 22.8
Statistical Analysis 1: Comparison: Brolucizumab 3 mg vs Aflibercept 2 mg; Test type: Other — Descriptive; Week 28; Bootstrap method; Difference - % = -0.3, 95% CI 2-sided [-6.4 to 5.8]
Statistical Analysis 2: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Other — Descriptive; Week 28; Bootstrap method; Difference - % = 4.6, 95% CI 2-sided [-1.3 to 11.0]
Statistical Analysis 3: Comparison: Brolucizumab 3 mg vs Aflibercept 2 mg; Test type: Other — Descriptive; Week 52; Bootstrap method; Difference - % = -4.2, 95% CI 2-sided [-10.2 to 2.2]
Statistical Analysis 4: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Other — Descriptive; Week 52; Bootstrap method; Difference - % = 3.9, 95% CI 2-sided [-2.2 to 10.5]
Statistical Analysis 5: Comparison: Brolucizumab 3 mg vs Aflibercept 2 mg; Test type: Other — Descriptive; Week 72; Bootstrap method; Difference - % = -9.2, 95% CI 2-sided [-15.5 to -2.8]
Statistical Analysis 6: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Other — Descriptive; Week 72; Bootstrap method; Difference - % = -2.3, 95% CI 2-sided [-8.4 to 4.4]
Statistical Analysis 7: Comparison: Brolucizumab 3 mg vs Aflibercept 2 mg; Test type: Other — Descriptive; Week 100; Bootstrap method; Difference - % = -7.7, 95% CI 2-sided [-14.0 to -1.6]
Statistical Analysis 8: Comparison: Brolucizumab 6 mg vs Aflibercept 2 mg; Test type: Other — Descriptive; Week 100; Bootstrap method; Difference - % = 0.4, 95% CI 2-sided [-5.7 to 6.8]

20. Secondary Outcome: Change From Baseline in Patient Reported Outcomes Visual Functioning Questionnaire-25 (VFQ-25) Total Scores up to Week 52 and Week 100 - Composite Score
Description: The National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) measures the influence of visual disability and visual symptoms on general health domains.
  The NEI VFQ-25 consists of a base set of 25 vision-targeted questions representing 11 vision-related constructs, plus an additional single-item general health rating question. All items are scored so that a high score represents better visual functioning. Each item is then converted to a 0 to 100 scale so that the lowest and highest possible scores are set at 0 and 100 points, respectively. A composite score is derived based on the average of the 11 subscales.
Time Frame: Baseline, Weeks 28, 52, 76, 100
Population: FAS - Observed
Measure: Mean (Standard Deviation); unit: overall scores
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 165 | 173 | 168
overall scores
  Week 28 | 5.5 (11.89) | 6.0 (14.27) | 7.8 (12.68)
  Week 52 (n = 151,148,157): number analyzed (Participants) | 151 | 148 | 157
  Week 52 (n = 151,148,157) | 4.6 (12.89) | 6.7 (13.24) | 8.5 (12.99)
  Week 76 (n = 133,138,143): number analyzed (Participants) | 133 | 138 | 143
  Week 76 (n = 133,138,143) | 6.7 (13.21) | 5.8 (14.50) | 7.1 (12.49)
  Week 100 (n=140,141,142): number analyzed (Participants) | 140 | 141 | 142
  Week 100 (n=140,141,142) | 6.6 (15.16) | 6.5 (14.41) | 6.2 (13.16)

21. Secondary Outcome: Change From Baseline in Patient Reported Outcomes Visual Functioning Questionnaire-25 (VFQ-25) Total Scores up to Week 52 and Week 100 - General Vision
Description: as for outcome 20
Time Frame: Baseline, Weeks 28, 52, 76, 100
Population: FAS - Observed
Measure: Mean (Standard Deviation); unit: overall scores
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 165 | 173 | 168
overall scores
  Week 28 | 7.8 (14.75) | 10.8 (18.11) | 11.3 (15.88)
  Week 52 (n = 151,148,157): number analyzed (Participants) | 151 | 148 | 157
  Week 52 (n = 151,148,157) | 6.6 (14.74) | 11.2 (17.18) | 10.7 (17.62)
  Week 76 (n = 133,138,143): number analyzed (Participants) | 133 | 138 | 143
  Week 76 (n = 133,138,143) | 7.5 (14.89) | 10.0 (17.80) | 11.7 (17.97)
  Week 100 (n=140,141,142): number analyzed (Participants) | 140 | 141 | 142
  Week 100 (n=140,141,142) | 10.4 (17.87) | 13.5 (17.97) | 11.5 (16.21)

22. Secondary Outcome: Change From Baseline in Patient Reported Outcomes Visual Functioning Questionnaire-25 (VFQ-25) Total Scores up to Week 52 and Week 100 - Ocular Pain
Description: as for outcome 20
Time Frame: Baseline, Weeks 28, 52, 76, 100
Population: FAS - Observed
Measure: Mean (Standard Deviation); unit: overall scores
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 165 | 173 | 168
overall scores
  Week 28 | 2.2 (21.02) | 2.4 (21.92) | 4.3 (23.61)
  Week 52 (n = 151,148,157): number analyzed (Participants) | 151 | 148 | 157
  Week 52 (n = 151,148,157) | 1.0 (19.55) | 4.9 (19.54) | 5.3 (22.16)
  Week 76 (n = 133,138,143): number analyzed (Participants) | 133 | 138 | 143
  Week 76 (n = 133,138,143) | 4.1 (19.75) | 2.1 (22.78) | 3.9 (21.72)
  Week 100 (n=140,141,142): number analyzed (Participants) | 140 | 141 | 142
  Week 100 (n=140,141,142) | 3.1 (19.90) | 3.1 (18.37) | 2.0 (19.73)

23. Secondary Outcome: Change From Baseline in Patient Reported Outcomes Visual Functioning Questionnaire-25 (VFQ-25) Total Scores up to Week 52 and Week 100 - Near Activities
Description: as for outcome 20
Time Frame: Baseline, Weeks 28, 52, 76, 100
Population: FAS - Observed
Measure: Mean (Standard Deviation); unit: overall scores
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 165 | 173 | 168
overall scores
  Week 28 | 8.4 (19.83) | 13.2 (24.93) | 13.7 (20.51)
  Week 52 (n = 151,148,157): number analyzed (Participants) | 151 | 148 | 157
  Week 52 (n = 151,148,157) | 8.1 (21.41) | 14.1 (24.17) | 13.4 (23.64)
  Week 76 (n = 133,138,143): number analyzed (Participants) | 133 | 138 | 143
  Week 76 (n = 133,138,143) | 11.7 (20.00) | 14.9 (23.35) | 12.4 (20.92)
  Week 100 (n=140,141,142): number analyzed (Participants) | 140 | 141 | 142
  Week 100 (n=140,141,142) | 11.6 (22.23) | 15.7 (22.01) | 10.4 (23.50)

24. Secondary Outcome: Change From Baseline in Patient Reported Outcomes Visual Functioning Questionnaire-25 (VFQ-25) Total Scores up to Week 52 and Week 100 - Distance Activities
Description: as for outcome 20
Time Frame: Baseline, Weeks 28, 52, 76, 100
Population: FAS - Observed
Measure: Mean (Standard Deviation); unit: overall scores
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 165 | 173 | 168
overall scores
  Week 28 | 6.0 (18.39) | 7.9 (21.58) | 9.0 (19.35)
  Week 52 (n = 151,148,157): number analyzed (Participants) | 151 | 148 | 157
  Week 52 (n = 151,148,157) | 4.2 (22.20) | 9.0 (19.42) | 9.9 (20.05)
  Week 76 (n = 133,138,143): number analyzed (Participants) | 133 | 138 | 143
  Week 76 (n = 133,138,143) | 8.3 (20.45) | 8.1 (19.20) | 7.0 (18.39)
  Week 100 (n=140,141,142): number analyzed (Participants) | 140 | 141 | 142
  Week 100 (n=140,141,142) | 6.4 (20.68) | 7.0 (19.24) | 6.7 (19.15)

25. Secondary Outcome: Change From Baseline in Patient Reported Outcomes Visual Functioning Questionnaire-25 (VFQ-25) Total Scores up to Week 52 and Week 100 - Social Functioning
Description: as for outcome 20
Time Frame: Baseline, Weeks 28, 52, 76, 100
Population: FAS - Observed
Measure: Mean (Standard Deviation); unit: overall scores
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 165 | 173 | 168
overall scores
  Week 28 | 2.7 (17.79) | 2.2 (18.00) | 3.9 (14.15)
  Week 52 (n = 151,148,157): number analyzed (Participants) | 151 | 148 | 157
  Week 52 (n = 151,148,157) | 3.1 (18.82) | 2.7 (17.53) | 3.8 (15.98)
  Week 76 (n = 133,138,143): number analyzed (Participants) | 133 | 138 | 143
  Week 76 (n = 133,138,143) | 3.6 (17.24) | 0.5 (18.95) | 1.7 (16.49)
  Week 100 (n=140,141,142): number analyzed (Participants) | 140 | 141 | 142
  Week 100 (n=140,141,142) | 2.5 (19.68) | 2.0 (21.82) | 1.4 (16.38)

26. Secondary Outcome: Change From Baseline in Patient Reported Outcomes Visual Functioning Questionnaire-25 (VFQ-25) Total Scores up to Week 52 and Week 100 - Mental Health
Description: as for outcome 20
Time Frame: Baseline, Weeks 28, 52, 76, 100
Population: FAS - Observed
Measure: Mean (Standard Deviation); unit: overall scores
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 165 | 173 | 168
overall scores
  Week 28 | 7.8 (20.63) | 8.2 (22.21) | 8.7 (19.71)
  Week 52 (n = 151,148,157): number analyzed (Participants) | 151 | 148 | 157
  Week 52 (n = 151,148,157) | 7.9 (22.93) | 9.6 (21.42) | 11.3 (21.34)
  Week 76 (n = 133,138,143): number analyzed (Participants) | 133 | 138 | 143
  Week 76 (n = 133,138,143) | 10.3 (21.07) | 11.5 (21.10) | 11.2 (20.93)
  Week 100 (n=140,141,142): number analyzed (Participants) | 140 | 141 | 142
  Week 100 (n=140,141,142) | 11.7 (25.28) | 9.4 (23.62) | 10.9 (22.22)

27. Secondary Outcome: Change From Baseline in Patient Reported Outcomes Visual Functioning Questionnaire-25 (VFQ-25) Total Scores up to Week 52 and Week 100 - Role Difficulties
Description: as for outcome 20
Time Frame: Baseline, Weeks 28, 52, 76, 100
Population: FAS - Observed
Measure: Mean (Standard Deviation); unit: overall scores
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 165 | 173 | 168
overall scores
  Week 28 | 8.0 (24.93) | 6.5 (26.81) | 9.4 (27.34)
  Week 52 (n = 151,148,157): number analyzed (Participants) | 151 | 148 | 157
  Week 52 (n = 151,148,157) | 6.9 (23.88) | 6.1 (29.11) | 11.3 (25.47)
  Week 76 (n = 133,138,143): number analyzed (Participants) | 133 | 138 | 143
  Week 76 (n = 133,138,143) | 9.9 (25.10) | 6.8 (29.48) | 7.4 (27.76)
  Week 100 (n=140,141,142): number analyzed (Participants) | 140 | 141 | 142
  Week 100 (n=140,141,142) | 9.3 (28.27) | 9.6 (28.88) | 6.9 (26.19)

28. Secondary Outcome: Change From Baseline in Patient Reported Outcomes Visual Functioning Questionnaire-25 (VFQ-25) Total Scores up to Week 52 and Week 100 - Dependency
Description: as for outcome 20
Time Frame: Baseline, Weeks 28, 52, 76, 100
Population: FAS - Observed
Measure: Mean (Standard Deviation); unit: overall scores
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 165 | 173 | 168
overall scores
  Week 28 | 6.3 (21.80) | 6.1 (25.16) | 7.1 (22.06)
  Week 52 (n = 151,148,157): number analyzed (Participants) | 151 | 148 | 157
  Week 52 (n = 151,148,157) | 3.8 (23.05) | 4.1 (25.36) | 9.0 (22.68)
  Week 76 (n = 133,138,143): number analyzed (Participants) | 133 | 138 | 143
  Week 76 (n = 133,138,143) | 5.2 (22.93) | 4.2 (25.56) | 6.8 (22.59)
  Week 100 (n=140,141,142): number analyzed (Participants) | 140 | 141 | 142
  Week 100 (n=140,141,142) | 5.5 (24.89) | 3.2 (25.79) | 5.6 (25.35)

29. Secondary Outcome: Change From Baseline in Patient Reported Outcomes Visual Functioning Questionnaire-25 (VFQ-25) Total Scores up to Week 52 and Week 100 - Driving
Description: as for outcome 20
Time Frame: Baseline, Weeks 28, 52, 76, 100
Population: FAS - Observed
Measure: Mean (Standard Deviation); unit: overall scores
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 108 | 107 | 100
overall scores
  Week 28 | 4.7 (16.40) | 1.9 (17.74) | 6.7 (15.06)
  Week 52 (n = 97,98,91): number analyzed (Participants) | 97 | 98 | 91
  Week 52 (n = 97,98,91) | 5.2 (16.51) | 3.6 (18.73) | 6.4 (17.64)
  Week 76 (n = 86,86,83): number analyzed (Participants) | 86 | 86 | 83
  Week 76 (n = 86,86,83) | 5.5 (16.09) | 2.9 (18.34) | 6.5 (19.13)
  Week 100 (n=86,86,81): number analyzed (Participants) | 86 | 86 | 81
  Week 100 (n=86,86,81) | 6.2 (16.58) | 4.3 (20.24) | 2.3 (18.84)

30. Secondary Outcome: Change From Baseline in Patient Reported Outcomes Visual Functioning Questionnaire-25 (VFQ-25) Total Scores up to Week 52 and Week 100 - Color Vision
Description: as for outcome 20
Time Frame: Baseline, Weeks 28, 52, 76, 100
Population: FAS - Observed
Measure: Mean (Standard Deviation); unit: overall scores
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 162 | 171 | 165
overall scores
  Week 28 | 2.6 (14.37) | 2.6 (18.20) | 1.8 (14.49)
  Week 52 (n = 148,147,152): number analyzed (Participants) | 148 | 147 | 152
  Week 52 (n = 148,147,152) | 2.0 (16.11) | 2.0 (12.59) | 1.6 (15.13)
  Week 76 (n = 131,137,140): number analyzed (Participants) | 131 | 137 | 140
  Week 76 (n = 131,137,140) | 1.7 (13.58) | 0.2 (17.01) | 0.2 (13.90)
  Week 100 (n=139,138,138): number analyzed (Participants) | 139 | 138 | 138
  Week 100 (n=139,138,138) | 2.0 (14.14) | 1.3 (15.79) | 0.5 (16.94)

31. Secondary Outcome: Change From Baseline in Patient Reported Outcomes Visual Functioning Questionnaire-25 (VFQ-25) Total Scores up to Week 52 and Week 100 - Peripheral Vision
Description: as for outcome 20
Time Frame: Baseline, Weeks 28, 52, 76, 100
Population: FAS - Observed
Measure: Mean (Standard Deviation); unit: overall scores
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 165 | 171 | 168
overall scores
  Week 28 | 3.6 (20.89) | 1.6 (22.05) | 9.2 (22.82)
  Week 52 (n = 151,148,156): number analyzed (Participants) | 151 | 148 | 156
  Week 52 (n = 151,148,156) | 1.3 (22.51) | 4.1 (22.97) | 8.5 (22.98)
  Week 76 (n = 133, 138, 143): number analyzed (Participants) | 133 | 138 | 143
  Week 76 (n = 133, 138, 143) | 5.6 (21.01) | 1.1 (24.33) | 7.3 (20.94)
  Week 100 (n=140, 140, 142): number analyzed (Participants) | 140 | 140 | 142
  Week 100 (n=140, 140, 142) | 3.4 (21.87) | -0.4 (24.36) | 6.3 (24.81)

32. Secondary Outcome: Change From Baseline in Patient Reported Outcomes Visual Functioning Questionnaire-25 (VFQ-25) Total Scores up to Week 52 and Week 100 - General Health Rating
Description: as for outcome 20
Time Frame: Baseline, Weeks 28, 52, 76, 100
Population: FAS - Observed
Measure: Mean (Standard Deviation); unit: overall scores
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 165 | 173 | 168
overall scores
  Week 28 | 0.9 (19.50) | 3.0 (22.10) | 6.1 (19.25)
  Week 52 (n = 151,148,157): number analyzed (Participants) | 151 | 148 | 157
  Week 52 (n = 151,148,157) | 4.3 (22.50) | 6.8 (22.32) | 6.8 (24.94)
  Week 76 (n = 133, 138, 143): number analyzed (Participants) | 133 | 138 | 143
  Week 76 (n = 133, 138, 143) | 2.3 (23.53) | 6.3 (24.18) | 8.2 (20.93)
  Week 100 (n=140, 141, 142): number analyzed (Participants) | 140 | 141 | 142
  Week 100 (n=140, 141, 142) | 2.3 (23.97) | 6.9 (23.55) | 8.8 (21.72)

33. Secondary Outcome: Ocular Adverse Events (AEs) (>=2% in Any Treatment Arm) by Preferred Term for the Study Eye
Time Frame: Adverse events were reported from first dose of study treatment until Week 96, plus 30 days post treatment, up to a maximum duration of 100 weeks.
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 190 | 189 | 187
Participants
  Number of subjects with at least one AE | 103 | 92 | 94
  Cataract | 17 | 16 | 13
  Conjunctival haemorrhage | 19 | 16 | 19
  Intraocular pressure increased | 14 | 11 | 3
  Vitreous detachment | 9 | 10 | 3
  Vitreous floaters | 7 | 10 | 6
  Diabetic retinal oedema | 12 | 9 | 4
  Conjunctivitis | 4 | 6 | 1
  Dry eye | 10 | 6 | 5
  Eye pain | 3 | 6 | 5
  Posterior capsule opacification | 3 | 6 | 3
  Eye irritation | 3 | 5 | 4
  Blepharitis | 3 | 4 | 4
  Keratitis | 0 | 4 | 3
  Vitreous haemorrhage | 2 | 4 | 3
  Punctate keratitis | 8 | 3 | 1
  Vision blurred | 6 | 3 | 1
  Visual acuity reduced | 7 | 3 | 9
  Iridocyclitis | 4 | 2 | 0
  Ocular hypertension | 4 | 2 | 2
  Uveitis | 4 | 2 | 0
  Corneal abrasion | 3 | 1 | 4
  Retinal exudates | 7 | 1 | 3
  Cataract subcapsular | 1 | 0 | 4
  Conjunctival hyperaemia | 4 | 0 | 1
  Vitreoretinal traction syndrome | 1 | 0 | 5

34. Secondary Outcome: Number of Subjects With Non-ocular Adverse Events (AEs) (>=2% in Any Treatment Arm)
Time Frame: as for outcome 33
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Brolucizumab 3 mg | Brolucizumab 6 mg | Aflibercept 2 mg
Number analyzed (Participants) | 190 | 189 | 187
Participants | 146 | 146 | 143

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until Week 96, plus 30 days post treatment, up to a maximum duration of 100 weeks.
Groups:
- Brolucizumab 3mg: Brolucizumab 3mg
- Brolucizumab 6mg: Brolucizumab 6mg
- Aflibercept 2mg: Aflibercept 2mg
- Overall: Overall
Arm/Group | Brolucizumab 3mg | Brolucizumab 6mg | Aflibercept 2mg | Overall
All-Cause Mortality (participants affected / at risk) | 4/190 | 8/189 | 7/187 | 19/566
Serious Adverse Events (participants affected / at risk) | 58/190 | 59/189 | 63/187 | 180/566
Other Adverse Events (participants affected / at risk) | 146/190 | 148/189 | 137/187 | 431/566
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab 3mg (N=190) | Brolucizumab 6mg (N=189) | Aflibercept 2mg (N=187) | Overall (N=566)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 1
Acute left ventricular failure (Cardiac disorders) | 0 | 0 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 2 | 3
Angina pectoris (Cardiac disorders) | 2 | 0 | 1 | 3
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 2 | 3
Atrioventricular block (Cardiac disorders) | 1 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1 | 0 | 2
Cardiac failure (Cardiac disorders) | 1 | 2 | 1 | 4
Cardiac failure chronic (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 5 | 2 | 5 | 12
Cardiorenal syndrome (Cardiac disorders) | 0 | 0 | 1 | 1
Cardiovascular disorder (Cardiac disorders) | 0 | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 2 | 3 | 6
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 1
Mitral valve disease mixed (Cardiac disorders) | 1 | 0 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 2 | 3 | 3 | 8
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 1
Goitre (Endocrine disorders) | 0 | 0 | 1 | 1
Amaurosis fugax - Fellow eye (Eye disorders) | 1 | 0 | 0 | 1
Cataract - Fellow eye (Eye disorders) | 0 | 3 | 4 | 7
Cataract - Study eye (Eye disorders) | 1 | 5 | 3 | 9
Conjunctival cyst - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Diabetic retinal oedema - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Diabetic retinopathy - Fellow eye (Eye disorders) | 0 | 0 | 1 | 1
Epiretinal membrane - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Glaucoma - Fellow eye (Eye disorders) | 0 | 0 | 1 | 1
Glaucoma - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Macular oedema - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Posterior capsule opacification - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Pterygium - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Retinal artery occlusion - Fellow eye (Eye disorders) | 1 | 0 | 0 | 1
Retinal artery occlusion - Study eye (Eye disorders) | 1 | 1 | 0 | 2
Retinal detachment - Study eye (Eye disorders) | 1 | 0 | 1 | 2
Retinal occlusive vasculitis - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Retinal vasculitis - Study eye (Eye disorders) | 2 | 0 | 0 | 2
Retinal vein thrombosis - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Uveitis - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Visual acuity reduced - Study eye (Eye disorders) | 0 | 0 | 1 | 1
Vitreous floaters - Study eye (Eye disorders) | 0 | 1 | 0 | 1
Vitreous haemorrhage - Fellow eye (Eye disorders) | 2 | 1 | 0 | 3
Vitritis - Study eye (Eye disorders) | 1 | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Proctitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Rectal polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Ulcerative gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Death (General disorders) | 0 | 1 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 2 | 2
Oedema peripheral (General disorders) | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1 | 2
Sudden death (General disorders) | 1 | 0 | 1 | 2
Bile duct stone (Hepatobiliary disorders) | 0 | 2 | 0 | 2
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Gallbladder disorder (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 1 | 1
Appendicitis (Infections and infestations) | 1 | 1 | 0 | 2
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 2 | 3 | 2 | 7
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 1 | 2
Cellulitis (Infections and infestations) | 2 | 1 | 2 | 5
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 1
Diabetic foot infection (Infections and infestations) | 2 | 1 | 0 | 3
Encephalitis (Infections and infestations) | 0 | 1 | 0 | 1
Endophthalmitis - Study eye (Infections and infestations) | 2 | 0 | 1 | 3
Fungal sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Gas gangrene (Infections and infestations) | 1 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1 | 0 | 1
Localised infection (Infections and infestations) | 1 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 2 | 3 | 6
Osteomyelitis acute (Infections and infestations) | 1 | 0 | 0 | 1
Periodontitis (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 2 | 1 | 4
Pneumonia fungal (Infections and infestations) | 1 | 0 | 0 | 1
Postoperative abscess (Infections and infestations) | 1 | 0 | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Sepsis (Infections and infestations) | 2 | 2 | 0 | 4
Septic shock (Infections and infestations) | 1 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 2
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Cataract operation complication - Fellow eye (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 2
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Laryngeal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 2
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Skin flap necrosis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Hepatitis C antibody positive (Investigations) | 0 | 0 | 1 | 1
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 1
Intraocular pressure increased - Study eye (Investigations) | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 3 | 0 | 3
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 0 | 0 | 2 | 2
Cerebral atrophy (Nervous system disorders) | 0 | 0 | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 1 | 2
Cerebrovascular accident (Nervous system disorders) | 3 | 4 | 4 | 11
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 1
Lacunar stroke (Nervous system disorders) | 0 | 0 | 1 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1 | 1
Optic neuritis - Study eye (Nervous system disorders) | 1 | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 1
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 2 | 2 | 5
Bladder pain (Renal and urinary disorders) | 0 | 1 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 1 | 0 | 2
Diabetic nephropathy (Renal and urinary disorders) | 1 | 1 | 1 | 3
End stage renal disease (Renal and urinary disorders) | 0 | 0 | 1 | 1
Nephropathy (Renal and urinary disorders) | 0 | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1 | 4 | 6
Urinary bladder rupture (Renal and urinary disorders) | 0 | 0 | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Prostatic disorder (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 4
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 3
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Accelerated hypertension (Vascular disorders) | 0 | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 1
Dry gangrene (Vascular disorders) | 1 | 0 | 0 | 1
Embolism venous (Vascular disorders) | 0 | 1 | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1 | 0 | 1
Haematoma (Vascular disorders) | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 2 | 0 | 0 | 2
Hypertensive crisis (Vascular disorders) | 0 | 2 | 1 | 3
Hypertensive emergency (Vascular disorders) | 0 | 1 | 0 | 1
Hypertensive urgency (Vascular disorders) | 0 | 0 | 2 | 2
Hypotension (Vascular disorders) | 1 | 0 | 1 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 2 | 0 | 2
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brolucizumab 3mg (N=190) | Brolucizumab 6mg (N=189) | Aflibercept 2mg (N=187) | Overall (N=566)
Anaemia (Blood and lymphatic system disorders) | 6 | 9 | 9 | 24
Atrial fibrillation (Cardiac disorders) | 8 | 1 | 1 | 10
Cardiac failure congestive (Cardiac disorders) | 2 | 4 | 3 | 9
Vertigo (Ear and labyrinth disorders) | 2 | 3 | 5 | 10
Blepharitis - Fellow eye (Eye disorders) | 4 | 5 | 4 | 13
Blepharitis - Study eye (Eye disorders) | 3 | 4 | 4 | 11
Cataract - Fellow eye (Eye disorders) | 11 | 12 | 5 | 28
Cataract - Study eye (Eye disorders) | 17 | 12 | 10 | 39
Cataract subcapsular - Study eye (Eye disorders) | 1 | 0 | 4 | 5
Conjunctival haemorrhage - Fellow eye (Eye disorders) | 2 | 5 | 7 | 14
Conjunctival haemorrhage - Study eye (Eye disorders) | 19 | 16 | 19 | 54
Conjunctival hyperaemia - Study eye (Eye disorders) | 4 | 0 | 1 | 5
Conjunctivitis allergic - Fellow eye (Eye disorders) | 3 | 2 | 4 | 9
Diabetic retinal oedema - Fellow eye (Eye disorders) | 17 | 12 | 12 | 41
Diabetic retinal oedema - Study eye (Eye disorders) | 12 | 9 | 4 | 25
Diabetic retinopathy - Fellow eye (Eye disorders) | 6 | 6 | 8 | 20
Dry eye - Fellow eye (Eye disorders) | 9 | 5 | 5 | 19
Dry eye - Study eye (Eye disorders) | 11 | 6 | 5 | 22
Eye irritation - Fellow eye (Eye disorders) | 0 | 6 | 2 | 8
Eye irritation - Study eye (Eye disorders) | 3 | 5 | 4 | 12
Eye pain - Fellow eye (Eye disorders) | 2 | 2 | 4 | 8
Eye pain - Study eye (Eye disorders) | 3 | 6 | 5 | 14
Iridocyclitis - Study eye (Eye disorders) | 4 | 2 | 0 | 6
Keratitis - Study eye (Eye disorders) | 0 | 4 | 3 | 7
Macular oedema - Fellow eye (Eye disorders) | 5 | 6 | 2 | 13
Ocular hypertension - Fellow eye (Eye disorders) | 2 | 5 | 2 | 9
Ocular hypertension - Study eye (Eye disorders) | 4 | 2 | 2 | 8
Posterior capsule opacification - Study eye (Eye disorders) | 3 | 5 | 3 | 11
Punctate keratitis - Study eye (Eye disorders) | 8 | 3 | 1 | 12
Retinal exudates - Fellow eye (Eye disorders) | 5 | 3 | 3 | 11
Retinal exudates - Study eye (Eye disorders) | 7 | 1 | 3 | 11
Retinal haemorrhage - Fellow eye (Eye disorders) | 5 | 2 | 1 | 8
Retinal haemorrhage - Study eye (Eye disorders) | 4 | 0 | 2 | 6
Vision blurred - Study eye (Eye disorders) | 6 | 3 | 1 | 10
Visual acuity reduced - Fellow eye (Eye disorders) | 4 | 3 | 3 | 10
Visual acuity reduced - Study eye (Eye disorders) | 7 | 3 | 8 | 18
Vitreoretinal traction syndrome - Study eye (Eye disorders) | 1 | 0 | 5 | 6
Vitreous detachment - Fellow eye (Eye disorders) | 5 | 5 | 4 | 14
Vitreous detachment - Study eye (Eye disorders) | 9 | 10 | 3 | 22
Vitreous floaters - Fellow eye (Eye disorders) | 7 | 5 | 5 | 17
Vitreous floaters - Study eye (Eye disorders) | 7 | 10 | 6 | 23
Vitreous haemorrhage - Fellow eye (Eye disorders) | 4 | 4 | 5 | 13
Vitreous haemorrhage - Study eye (Eye disorders) | 2 | 4 | 3 | 9
Constipation (Gastrointestinal disorders) | 4 | 4 | 5 | 13
Diarrhoea (Gastrointestinal disorders) | 5 | 10 | 6 | 21
Nausea (Gastrointestinal disorders) | 2 | 5 | 3 | 10
Vomiting (Gastrointestinal disorders) | 5 | 7 | 2 | 14
Oedema peripheral (General disorders) | 4 | 5 | 5 | 14
Pyrexia (General disorders) | 1 | 8 | 3 | 12
Seasonal allergy (Immune system disorders) | 2 | 4 | 4 | 10
Bronchitis (Infections and infestations) | 5 | 5 | 4 | 14
COVID-19 (Infections and infestations) | 8 | 7 | 7 | 22
Cellulitis (Infections and infestations) | 0 | 2 | 4 | 6
Conjunctivitis - Fellow eye (Infections and infestations) | 3 | 6 | 4 | 13
Conjunctivitis - Study eye (Infections and infestations) | 4 | 6 | 1 | 11
Ear infection (Infections and infestations) | 4 | 0 | 2 | 6
Herpes zoster (Infections and infestations) | 5 | 0 | 0 | 5
Influenza (Infections and infestations) | 6 | 8 | 7 | 21
Lower respiratory tract infection (Infections and infestations) | 4 | 1 | 0 | 5
Nasopharyngitis (Infections and infestations) | 20 | 18 | 16 | 54
Pneumonia (Infections and infestations) | 3 | 4 | 4 | 11
Sinusitis (Infections and infestations) | 4 | 5 | 4 | 13
Tooth infection (Infections and infestations) | 1 | 0 | 4 | 5
Upper respiratory tract infection (Infections and infestations) | 6 | 5 | 5 | 16
Urinary tract infection (Infections and infestations) | 17 | 20 | 8 | 45
Corneal abrasion - Study eye (Injury, poisoning and procedural complications) | 3 | 1 | 4 | 8
Fall (Injury, poisoning and procedural complications) | 5 | 5 | 2 | 12
Limb injury (Injury, poisoning and procedural complications) | 4 | 1 | 1 | 6
Blood glucose increased (Investigations) | 2 | 4 | 1 | 7
Blood pressure increased (Investigations) | 6 | 4 | 3 | 13
Glucose urine present (Investigations) | 1 | 4 | 2 | 7
Glycosylated haemoglobin increased (Investigations) | 4 | 1 | 4 | 9
Intraocular pressure increased - Fellow eye (Investigations) | 5 | 0 | 3 | 8
Intraocular pressure increased - Study eye (Investigations) | 14 | 11 | 3 | 28
Dehydration (Metabolism and nutrition disorders) | 2 | 6 | 0 | 8
Diabetes mellitus (Metabolism and nutrition disorders) | 7 | 4 | 7 | 18
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 4 | 3 | 3 | 10
Dyslipidaemia (Metabolism and nutrition disorders) | 2 | 4 | 2 | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 4 | 1 | 7
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 | 6 | 3 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 6 | 5 | 23
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 6 | 15
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2 | 6
Dizziness (Nervous system disorders) | 5 | 4 | 3 | 12
Headache (Nervous system disorders) | 3 | 10 | 3 | 16
Migraine (Nervous system disorders) | 1 | 2 | 5 | 8
Depression (Psychiatric disorders) | 0 | 4 | 3 | 7
Acute kidney injury (Renal and urinary disorders) | 1 | 4 | 3 | 8
Chronic kidney disease (Renal and urinary disorders) | 1 | 7 | 7 | 15
Renal failure (Renal and urinary disorders) | 5 | 2 | 3 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 11 | 10 | 28
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 2 | 8
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 | 4 | 2 | 10
Hypertension (Vascular disorders) | 22 | 21 | 24 | 67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT03481634/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-26): https://cdn.clinicaltrials.gov/large-docs/34/NCT03481634/SAP_002.pdf